CLINICAL TRIAL: NCT03020446
Title: Effectiveness of Sorbion in the Treatment of Venous Leg Ulcers The Protocol Elements
Acronym: Sorbion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Provider of product no longer wished to continue with site. No data available.
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sorbion Study
Record Dates: First submitted 2015-10-07; First posted 2017-01-13 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Venous Wound Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorbion dressing to venous leg ulcer (Experimental): any venous leg ulcer will receive sorbion dressing weekly for 4 weeks than wound will be assessed
  Interventions: Device: Sorbion Dressing

INTERVENTIONS:
Device: Sorbion Dressing — Sorbion dressing will be placed on venous leg ulcer and changed weekly for 4 weeks
  Other Names: Sorbion Sachet sorbion sana

SUMMARY:
To follow the effectiveness of Sorbion Dressing in the treatment of highly exuding venous leg ulcers.

DETAILED DESCRIPTION:
Wounds will be assessed for inclusion into the study, digital images of the wound will be taken, wound will be cleansed, a sorbion dressing will be placed on wound and a cover dressing with be used to keep in place. The wound will be assessed and a dressing change will take place weekly for 4 weeks. At the final visit a final wound evaluation will be done.

ELIGIBILITY:
Inclusion Criteria:

* venous leg ulcer

Exclusion Criteria:

* pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toledo Medical Center, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorbion Dressing to Venous Leg Ulcer
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sorbion Dressing to Venous Leg Ulcer
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 67 [62 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Wound Size
Description: decreased wound bed measured in centimeters
Time Frame: 4 weeks
Population: Study was terminated
Arm/Group | Sorbion Dressing to Venous Leg Ulcer
Number analyzed (Participants) | 0

2. Secondary Outcome: Wound Maceration
Description: visual assessment of decreased wound maceration
Time Frame: 4 weeks
Population: Study was termininated
Arm/Group | Sorbion Dressing to Venous Leg Ulcer
Number analyzed (Participants) | 0

3. Secondary Outcome: Wound Necrosis
Description: visual assessment of decreased wound necrosis
Time Frame: 4 weeks
Population: Study was terminated
Arm/Group | Sorbion Dressing to Venous Leg Ulcer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sorbion Dressing to Venous Leg Ulcer
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes